CLINICAL TRIAL: NCT00519805
Title: FRAGMATIC - A Randomised Phase III Clinical Trial Investigating the Effect of FRAGMin Added to Standard Therapy In Patients With Lung Cancer
Brief Title: Dalteparin in Preventing Blood Clots in Patients With Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Velindre NHS Trust (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000561532; WCTU-FRAGMATIC; Velindre-FRAGMATIC; WCTU-02; EU-20753; PFIZER-WCTU-02; EUDRACT-2005-002438-37; ISRCTN80812769
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2008-03

CONDITIONS: Lung Cancer; Thromboembolism
Keywords: thromboembolism; extensive stage small cell lung cancer; limited stage small cell lung cancer; stage IV non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Thromboembolism; Carcinoma, Non-Small-Cell Lung | interventions — Dalteparin

INTERVENTIONS:
Drug: dalteparin
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Anticoagulants, such as dalteparin, may help prevent blood clots from forming in patients with lung cancer. It is not yet known whether dalteparin is effective in preventing blood clots in patients with lung cancer.

PURPOSE: This randomized phase III trial is studying how well dalteparin works in preventing blood clots in patients with lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the addition of dalteparin results in improved survival.

Secondary

* Determine venous thrombotic event-free survival and metastasis-free survival.
* Determine serious adverse events in patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the quality of life, breathlessness, anxiety, and depression in patients treated with this drug.
* Determine the cost effectiveness and cost utility of this drug.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients receive anticancer treatment considered appropriate by the local medical team.
* Arm II: Patients receive anticancer treatment considered appropriate by the local medical team. Beginning before the start of the first definitive anticancer treatment, patients receive dalteparin subcutaneously daily for up to 24 weeks.

Quality of life, anxiety, depression, and dyspnea are assessed at baseline, at 12 and 24 weeks, and then at 9 and 12 months.

After completion of therapy, patients are followed at 9 months, 1 year, and then every 6 months for at least 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathological or cytological diagnosis of primary bronchial carcinoma (small cell or non-small cell lung cancer) within the past 6 weeks
* No other intrathoracic tumors (e.g., carcinoid tumor, mesothelioma, lymphoma, or lung metastases from another primary site)
* No clinically apparent brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 150 µmol/L
* Willing and able to self-administer dalteparin by daily subcutaneous injection or have it administered by a caregiver
* Not pregnant or nursing
* Fertile female patients must use effective contraception (if sexually active)
* No hemorrhagic stroke within the past 3 months
* No known bleeding disorder
* No hemoptysis of CTC ≥ grade 2 (i.e., symptomatic hemoptysis requiring medical intervention)
* No central venous catheter requiring the use of thromboprophylaxis
* No known hypersensitivity to dalteparin, heparin, or other low molecular weight heparins (e.g., history of confirmed or suspected immunologically mediated heparin-induced thrombocytopenia; acute gastroduodenal ulcer; or subacute endocarditis)
* No prior illness likely to interfere with study treatment or comparisons

PRIOR CONCURRENT THERAPY:

* No prior treatment likely to interfere with study treatment or comparisons
* More than 12 months since prior and no concurrent therapeutic anticoagulation
* No concurrent ketorolac (Toradol®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2007-08; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Venous thrombotic event-free survival
Serious adverse events
Metastasis-free survival
Toxicity
Quality of life as measured by EQ-5D
Breathlessness (dyspnea) as measured by the Cancer Dyspnea Scale
Anxiety and depression as measured by the Hospital Anxiety and Depression Scale
Cost effectiveness
Cost utility

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Macbeth, MD, Study Chair — Velindre NHS Trust
Locations (60):
- United Kingdom (60):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Furness General Hospital, Barrow in Furness, England
  - Royal Blackburn Hospital, Blackburn, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Burnley General Hospital, Burnley, England
  - Queen's Hospital, Burton-on-Trent, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Walsgrave Hospital, Coventry, England
  - Darlington Memorial, Darlington, England
  - Derbyshire Royal Infirmary, Derby, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Dorset County Hospital, Dorchester, England
  - Russells Hall Hospital, Dudley, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Wycombe General Hospital, High Wycombe, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Whipps Cross Hospital, London, England
  - Saint Bartholomew's Hospital, London, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - Whittington Hospital, London, England
  - University College Hospital, London, England
  - UCL Cancer Institute, London, England
  - Luton and Dunstable Hospital, Luton, England
  - James Cook University Hospital, Middlesbrough, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - James Paget Hospital, Norfolk, England
  - North Tyneside Hospital, North Shields, England
  - Friarage Hospital, North Yorks, England
  - Northampton General Hospital, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital, Nottingham, England
  - George Eliot Hospital, Nuneaton, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Scarborough General Hospital, Scarborough, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - South Tyneside District Hospital, South Shields, England
  - Staffordshire General Hospital, Stafford, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Royal Marsden - Surrey, Sutton, England
  - South Warwickshire Hospital, Warwick, Warwickshire, England
  - Weston General Hospital, Weston-super-Mare, England
  - New Cross Hospital, Wolverhampton, England
  - Yeovil District Hospital, Yeovil, England
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Llandough Hospital, Llandough, Wales
  - Royal Glamorgan Hospital, Llantrisant, Wales
  - Prince Charles Hospital, Mid Glamorgan, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales

REFERENCES:
- [Result] Griffiths GO, Burns S, Noble SI, Macbeth FR, Cohen D, Maughan TS. FRAGMATIC: a randomised phase III clinical trial investigating the effect of fragmin added to standard therapy in patients with lung cancer. BMC Cancer. 2009 Oct 6;9:355. doi: 10.1186/1471-2407-9-355. PMID 19807917
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539